CLINICAL TRIAL: NCT03128242
Title: An Eye-tracking Study to Investigate Oxytocin's Effect on Attentional Bias Training
Brief Title: Oxytocin's Effect on Attention Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-32
Record Dates: First submitted 2017-04-17; First posted 2017-04-25 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: oxytocin; attention bias; attention training; eye-tracking
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxytocin group (Experimental): oxytocin treatment
  Interventions: Drug: Oxytocin
- placebo group (Placebo Comparator): placebo treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Oxytocin — intranasal administration of oxytocin (24IU)
  Arms: oxytocin group
Drug: placebo — intranasal administration of placebo (24IU)
  Arms: placebo group

SUMMARY:
This study aims to investigate oxytocin's effect on attentional bias training. Healthy participants will undergo a dot-probe task-based training to direct their attention away from negative stimuli (as compared to neutral). Effects of the training will be assessed using an eye-tracking anti-saccade task.

DETAILED DESCRIPTION:
In this study, a dot-probe task will be used to examine if subjects show an attentional bias towards negative stimuli and whether the bias can be modified using a subsequent attentional bias training. During this training participants learn to direct their attention away from threatening stimuli. In a between-subject placebo controlled design participants will receive either intranasal oxytocin or placebo before the training to examine whether oxytocin could facilitate the effects of the attention training. Effects of the training and of oxytocin on the training will be assessed by means of an eye-tracking anti-saccade task. Based on previous studies showing the strongest effects of threat-attentional bias training in high anxious subjects, the study will recruit participants with an elevated trait anxiety.

ELIGIBILITY:
Inclusion Criteria:

* male participants with elevated trait anxiety (> 45 scores as assessed with the State and Trait Anxiety Inventory, Spielberger, 1983)
* without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury
* medical or psychiatric illness
* smoking or drinking 24 hours before the experiment

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2016-11-25 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Reaction time (RT) difference - oxytocin effects | Before drug administration (pre-treatment baseline) and 55 minutes after drug administration
  Difference before and after oxytocin administration: reaction time to negative and neutral stimuli in the dot-probe task
Reaction time (RT) difference - training effects | Before drug administration - 55-90 minutes after drug administration
  Difference before and after training: reaction time to negative and neutral stimuli in the dot-probe task
Saccade latency difference - training effects | Before drug administration - 55-90 minutes after drug administration
  Difference before and after training in saccade latency in the anti-saccade task

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Becker, Dr., Principal Investigator — School of Life Science and Technology, University of Electronic Science and Technology of China
Locations (1):
- School of Life Science and Technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China